CLINICAL TRIAL: NCT04231617
Title: The Hemodynamic Effects of CGRP After Glibenclamide Administration in a Randomized Double-blind Cross-over Placebo-controlled Study With Healthy Volunteers
Brief Title: The Hemodynamic Effects of CGRP After Glibenclamide Administration in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Mohammad Al-Mahdi Al-Karagholi, MD, PhD student, Principal investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: H-19065735
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Hemodynamics of Cranial Arteries; Headache; Cerebral Blood Flow
MeSH Terms: conditions — Headache | interventions — Glyburide

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, cross-over, placebo-controlled design in healthy volunteers.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGRP and glibenclamide (Active Comparator): Participants will recieve CGRP infusion after glibenclamide/placebo administration
  Interventions: Drug: glibenclamide; Drug: CGRP infusion
- CGRP and placebo (Active Comparator): Participants will recieve CGRP infusion after glibenclamide/placebo administration
  Interventions: Drug: CGRP infusion; Drug: Placebo

INTERVENTIONS:
Drug: glibenclamide — Oral administration of glibenclamide or placebo. To investigate the role of CGRP on cranial arteries in healthy volunteers after glibenclamide/placebo administration .
  Arms: CGRP and glibenclamide
Drug: CGRP infusion — CGRP infusion
Drug: Placebo — placebo
  Arms: CGRP and placebo

SUMMARY:
To investigate the hemodynamic effects of CGRP after glibenclamide administration.

DETAILED DESCRIPTION:
20 healthy participants will randomly be allocated to receive CGRP infusion followed by glibenclamide or placebo on two different days.

The aim of the study is to investigate the vascular effect of CGRP after glibenclamide administration.

Repeated measurements covering the arteria radialis (RA), superficiel temporal artery (STA) and middle cerebral artery (MCA) before and after glibenclamide/placebo administration and CGRP infusion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of both sexes.
* 18-60 years.
* 50-100 kg.
* Women of childbearing potential must use adequate contraception

Exclusion Criteria:

* A history of serious somatic disease
* Migraine or any other type of headache (except episodic tension-type headache less than once a month)
* Daily intake of any medication except contraceptives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Changes in the arterial radialis (RA), superficiel temporal artery (STA) and middle cerebral artery (MCA) | Time of measurements is baseline and repeatedly every 20 min for 240 min.
  Repeated measurements covering the diameter of RA , STA and MCA before and after glibenclamide/placebo administration and CGRP infusion measured by centimeter (cm)

SECONDARY OUTCOMES:
Headache | Time of headache measurements is from before (-20 min) and after (12 hours) glibenclamide/placebo administration.
  Headache intensity will be recorded by numerical rating scale (NRS) from 0 to 10 (0, no headache; 1, a feeling of pressure; 10, worst imaginable headache).

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Danish headache center, Glostrup Municipality, Copenhagen
  - Mohammad Al-Mahdi Al-Karagholi, København S, Danmark